CLINICAL TRIAL: NCT06582966
Title: Weekly Doxycycline DOT for STI Prevention Among Cisgender Women Taking HIV PrEP in Kisumu, Kenya
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Jared Baeten, Professor: Global Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00019944; 5R01AI145971-04 (NIH)
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: STI
Keywords: STI
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: Open label, single-arm, pilot study of 60 cisgender women taking HIV PrEP in Kisumu, Kenya will be given doxycycline 200 mg orally once weekly with clinical follow-up including quarterly STI testing and treatment for six months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DoxyDOT single arm (Other): Open label, single-arm, pilot study of 60 cisgender women taking HIV PrEP in Kisumu, Kenya will be given doxycycline 200 mg orally once weekly with clinical follow-up including quarterly STI testing and treatment for six months.
  Interventions: Drug: Doxycyclin

INTERVENTIONS:
Drug: Doxycyclin — Open label, single-arm, pilot study of 60 cisgender women taking HIV PrEP in Kisumu, Kenya will be given doxycycline 200 mg orally once weekly with clinical follow-up including quarterly STI testing and treatment for six months.

SUMMARY:
The first study of doxycycline postexposure prophylaxis for cisgender women did not reduce incident STIs likely due to low use of doxycycline. Researchers will conduct a pilot study of once-weekly doxyxycline to prevent bacterial STIs among Kenyan cisgender women using PrEP for HIV prevention.

DETAILED DESCRIPTION:
A study evaluating doxycycline prophylaxis to prevent sexually transmitted infections (STIs) in PrEP-taking African women, who are a priority population for STI prevention, given their high risk and engagement in longitudinal prevention services. The primary study objective is to assess the acceptability of once weekly doxycycline prophylaxis and assess persistence in once weekly doxycycline delivered as directly observed therapy (DOT). STI prophylaxis carries substantial potential benefits but also important potential risks, and we have framed our work as capturing key data to inform this question. Researchers hypothesize that weekly doxycycline will substantially reduce the incidence of curable STIs, particularly C. trachomatis, the most common bacterial STI and the one responsible for greatest morbidity.

Researchers' secondary study objectives are to evaluate the impact on incidence rate of STIs in women given once-weekly doxycycline DOT in comparison with data collected among participants assigned to received standard of care in recently completed dPEP Kenya study as well as to assess tolerability of once weekly doxycycline prophylaxis. Researchers will collect samples for future doxycycline hair drug level testing, antibiotic resistance testing, and microbiome evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent
2. Age 18-30 years
3. Female sex assigned at birth
4. HIV-seronegative, according to national HIV testing algorithm
5. Has a current prescription for PrEP, > 1 month, according to the national guidelines of Kenya

Exclusion Criteria:

1. Pregnant
2. Breastfeeding a child
3. Allergy to tetracycline class
4. Current medications which may impact doxycycline metabolism or that are contraindicated with doxycycline, as per the prescribing information. These include systemic retinoids, barbiturates, carbamazepine, phenytoin, and warfarin.
5. Active, clinically significant medical or psychiatric conditions that would interfere with study participation, at the discretion of the site investigator or designee.
6. Prior enrollment in The dPEP Kenya Study

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — cis-gender women
Enrollment: 60 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
doxyPEP DOT adherence | 6 months
  Confirmation of weekly doxyPEP DOT dosing each week will be recorded on weekly CRFs and quarterly surveys on acceptability will be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Baeten, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- Kenya Medical Research Institute -KEMRI, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No